CLINICAL TRIAL: NCT07243964
Title: Multi-Omics-Based Prediction of Allograft Dysfunction After Lung Transplantation: A Prospective, Multicenter Cohort Study
Brief Title: Multi-Omics-Based Prediction of Allograft Dysfunction After Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: Chang Chen (Other)
Responsible Party: Sponsor-Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Other Study IDs: L25-802
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: longitudinal changes in multi-omics profiling of peripheral blood — This study investigates the associations between longitudinal changes in multi-omics profiling of peripheral blood-including cell-free DNA, single-cell transcriptomics, proteomics, and metabolomics-and the development of acute lung allograft dysfunction(ALAD) and chronic lung allograft dysfunction(CLAD) in lung transplant recipients at various postoperative time points.

SUMMARY:
By establishing a prospective, multicenter lung transplantation clinical cohort, this study aims to systematically evaluate the utility of cfDNA fragmentomics, peripheral blood single-cell sequencing, and proteomics in monitoring and predicting graft dysfunction after lung transplantation, and to develop a multi-omics predictive model for early identification, dynamic monitoring, and mechanistic investigation of acute lung allograft dysfunction (ALAD) and chronic lung allograft dysfunction (CLAD).

DETAILED DESCRIPTION:
ALAD predominantly occurs in the early post-transplant period. This project aims to establish a systematic framework for monitoring and predicting post-lung transplant dysfunction, with a specific focus on acute lung allograft dysfunction (ALAD) and its progression to chronic lung allograft dysfunction (CLAD). We plan to conduct a prospective, multicenter clinical cohort study, longitudinally collecting peripheral blood and bronchoalveolar lavage fluid (BALF) samples from transplant recipients at various time points. By integrating multi-omics technologies-including cfDNA fragmentomics, peripheral blood single-cell sequencing, and proteomic mass spectrometry-with pulmonary function (FEV1) and clinicopathological data, we seek to delineate the dynamic landscape of post-lung transplant dysfunction. Compared to previous studies that relied on single indicators or one-time measurements, this project is distinguished by several key features: Firstly, the use of cfDNA fragmentomic characteristics to infer tissue origin, enabling highly specific detection of graft injury without requiring donor genotype information. Secondly, the integration of single-cell transcriptomics to comprehensively analyze the dynamics of peripheral immune cell subsets, providing a basis for early immunological warning of dysfunction. Thirdly, the application of proteomics to reveal expression levels, post-translational modifications, and protein-protein interactions in plasma samples. Fourthly, the construction of a multi-dimensional integrated model incorporating blood, BALF, and pulmonary function data, with the goal of establishing a generalizable early warning system. Through this research, we aim not only to enhance the early identification and intervention of ALAD but also to lay the foundation for elucidating the molecular mechanisms underlying CLAD development and exploring potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients aged ≥18 years undergoing single or double lung transplantation;
2. Postoperative recipients capable of understanding and providing written informed consent, and willing to comply with scheduled follow-ups and sample collections as required by the study;
3. Postoperative recipients clinically assessed as stable and eligible for routine follow-up and hematological examinations;
4. Recipients able to undergo dynamic pulmonary function monitoring during follow-up;
5. No planned participation in other interventional trials during the study period that may impact immune function or pulmonary function;
6. Retransplant patients will be considered as a new transplant event and may be included in the analysis.

Exclusion Criteria:

1. History of active malignancy or presence of untreated malignancy within 5 years prior to transplantation;
2. Presence of active systemic infection or significant immune rejection;
3. Female patients who are pregnant or lactating;
4. Any other condition deemed by the investigator to be inappropriate for inclusion .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recipients undergoing single or double lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ALAD | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD,PHD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No